CLINICAL TRIAL: NCT05544123
Title: A Multi-center, Observational Study to Describe the Treatment Situation of Chinese County Population With HER2+ & HR+/HER2- Breast Cancer
Brief Title: The Treatment Situation of Chinese County Population With Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Xinxiang Medical College (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: ESR-21-21505
Record Dates: First submitted 2022-09-09; First posted 2022-09-16 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer; Breast Carcinoma; Breast Tumor
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort 1 HER2+ EBC: newly diagnosed or completed definitive breast surgery
  Interventions: Other: pathological stage
- Cohort 2 HR+ HER2- EBC: newly diagnosed or completed definitive breast surgery
  Interventions: Other: pathological stage
- Cohort 3 HER2+ ABC: De novo or relapsed from adjuvant therapy
  Interventions: Other: pathological stage
- Cohort 4 HR+ HER2- ABC: De novo or relapsed from adjuvant therapy
  Interventions: Other: pathological stage

INTERVENTIONS:
Other: pathological stage — breast cancer molecular subtyping and pathological TNM stage

SUMMARY:
The study is a multi-center, non-interventional, prospective observational study which enrols 2500 breast cancer patients from China county area. The purpose of this study is to be aware of the real-world data of the current breast cancer diagnosis and treatment model in the county. It aims to understand the gap between the county and the SOC in the diagnosis and treatment.

DETAILED DESCRIPTION:
The study is a multi-center, non-interventional, prospective observational study which enrols 2500 breast cancer patients from China county area. The patients will be divided into four cohorts by HR/HER2 status and early/late stage without prespecified minimum or maximum limit of patient number for each cohort.

The potential study subjects will be identified by the investigators by face-to-face visit. During this process approximately 2500 subjects will be enrolled in 1 year. All subjects will be sign informed consent and recorded for demographic characteristics, medical history, treatment history, treatment hospital, pathologic diagnosis, receptor status, therapeutic regimen, etc at the beginning of enrollment. Normally, there will be 4 visits for EBC and 6 visits for ABC in hospitals during yearlong follow-up period. All visits are according to the standard frequency of clinical follow-up. If the patient does not come to the hospital for follow-up on a regular basis, we will follow-up by telephone inquiries, etc.The potential study subjects will be identified by the investigators by face-to-face visit. During this process approximately 2500 subjects will be enrolled in 1 year. All subjects will be sign informed consent and recorded for demographic characteristics, medical history, treatment history, treatment hospital, pathologic diagnosis, receptor status, therapeutic regimen, etc at the beginning of enrollment. Normally, there will be 4 visits for EBC and 6 visits for ABC in hospitals during yearlong follow-up period. All visits are according to the standard frequency of clinical follow-up. If the patient does not come to the hospital for follow-up on a regular basis, we will follow-up by telephone inquiries, etc.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1

* Age ≥ 18 years at the time of enrollment
* Histologically confirmed HER2+ breast cancer
* Newly diagnosed or completed definitive early breast surgery
* Complete medical history information

Cohort 2

* Age ≥ 18 years at the time of enrollment
* Histologically confirmed HR+ HER2- breast cancer
* Newly diagnosed or completed definitive early breast surgery
* Complete medical history information

Cohort 3

* Age ≥ 18 years at the time of enrollment
* Histologically confirmed HER2+ breast cancer
* De Novo or recurrent metastatic breast cancer
* Complete medical history information

Cohort 4

* Age ≥ 18 years at the time of enrollment
* Histologically confirmed HR+ HER2- breast cancer
* De Novo or recurrent metastatic breast cancer
* Complete medical history information

Exclusion Criteria:

Cohort 1

* Participated in other Intervention drug clinical trials within 4 weeks before admission Cohort 2
* Participated in other Intervention drug clinical trials within 4 weeks before admission Cohort 3
* Patients with HER2 + advanced breast cancer who have received more than 2 lines of therapy
* Participated in other Intervention drug clinical trials within 4 weeks before admission Cohort 4
* Patients with HR+ HER2- advanced breast cancer who have received more than 2 lines of therapy
* Participated in other Intervention drug clinical trials within 4 weeks before admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 2500 breast cancer patients will be recruited in this study. The entire subjects are spread over 13 Provinces (Henan province, Hebei province, Hunan Province etc.) and 2 autonomous regions (Inner Mongolia Autonomous Region and Guangxi Zhuang Autonomous Region). In order to acquire adequate treatment patterns choices in China county area. Data collection and analysis are needed in the corresponding population.
  Data collection and analysis are needed in the corresponding population. The entire subjects contain in this study are spread over 13 Provinces (Henan province, Hebei province, Hunan Province etc.) and 2 autonomous regions (Inner Mongolia Autonomous Region and Guangxi Zhuang Autonomous Region).
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2022-09-29 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
the treatment pattern in HER2+, and HR+HER2- early and advanced breast cancer patients in county in each cohort | 1 year
  Different treatment patterns in each cohort

SECONDARY OUTCOMES:
the referral behavior in county | 1 year
  To describe the referral behavior in county (Among all patients)
he relationship between recurrent risk and OFS, chemotherapy and OFS | 1 year
  To explore the relationship between recurrent risk and OFS, chemotherapy and OFS
the duration of medical OFS in early breast cancer | 1 year
  To explore the duration of medical OFS in early breast cancer
the duration of anti-HER2 therapy in advanced breast cancer | 1 year
  To explore the duration of anti-HER2 therapy in advanced breast cancer

OTHER OUTCOMES:
Proportion of re-biopsy of recurrent/metastatic disease | 1 year
  Proportion of re-biopsy of recurrent/metastatic disease
Rate of HER2 testing in county | 1 year
  Rate of HER2 testing in county (IHC and FISH) (Among all patients)
Percentage of Her-2 low expression among HR+HER2- early and advanced breast cancer (Cohort 2 and Cohort 4) | 1 year
  Percentage of Her-2 low expression among HR+HER2- early and advanced breast cancer (Cohort 2 and Cohort 4)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - 路平, Xinxiang, Henan

IPD SHARING:
Plan to Share IPD: No